CLINICAL TRIAL: NCT06572579
Title: Safety and Effectiveness of Ultrasound-guided Pharmacopuncture for Spinal Diseases: A Pilot Registry
Brief Title: A Pilot Registry for Ultrasound-guided Pharmacopuncture
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2024-04
Record Dates: First submitted 2024-07-22; First posted 2024-08-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-09

CONDITIONS: Neck Pain; Back Pain
MeSH Terms: conditions — Neck Pain; Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ultrasound-guided pharmacopuncture group: Patients diagnosed with spinal disorders who have undergone ultrasound-guided pharmacopuncture treatment
  Interventions: Procedure: Ultrasound-guided pharmacopuncture treatment

INTERVENTIONS:
Procedure: Ultrasound-guided pharmacopuncture treatment — Pharmacopuncture treatment using ultrasound-guidance

SUMMARY:
A pilot study of prospective resigstry to evaluate the safety and efficacy of ultrasound-guided pharmacopuncture for spinal disorders

DETAILED DESCRIPTION:
This study aims to evaluate the safety and efficacy of ultrasound-guided pharmacopuncture by collecting information on adverse reactions, efficacy assessment variables, and treatment methods from patients diagnosed with spinal disorders who have undergone ultrasound-guided pharmacopuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals diagnosed with spinal disorders (M code and S code based on KCD criteria)
2. Outpatients scheduled for ultrasound-guided pharmacopuncture treatment
3. Individuals aged 19 years or older and under 70 years
4. Individuals who agree to participate in the clinical study and voluntarily sign the consent form

Exclusion Criteria:

1. Individuals who are unable to complete the consent form
2. Individuals who are deemed unsuitable for participation in the clinical study by the researcher

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with spinal disorders who have undergone ultrasound-guided pharmacopuncture treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Adverse Event | Treatment visits up to 12 weeks, and Week 2, 4, 8, 12 follow-ups
  Adverse events assessment

SECONDARY OUTCOMES:
Spinal pain numeric rating scale | Week 0, Treatment visits up to 12 weeks, and Week 2, 4, 8, 12 follow-ups
  Spinal pain numeric rating scale
Disability index | Week 0, 2, 4, 8, 12
  Neck disability index or Oswestry Disability Index
EQ-5D-5L | Week 0, 2, 4, 8, 12
  Quality of life using EQ-5D-5L
Patient satisfaction | Week 4
  Patient satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Dr, Study Director — Jaseng Medical Foundation
Locations (3):
- South Korea (3):
  - Jaseng Hospital of Korean medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Daejeon Jaseng Hospital of Korean medicine, Daejeon, Seo-gu

IPD SHARING:
Plan to Share IPD: No